CLINICAL TRIAL: NCT03151967
Title: Lactobacillus Probiotic for Prevention of UTI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ann Stapleton, Professor, Medicine, Infectious Diseases, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00000160; 1R01DK088830-01A1 (NIH)
Record Dates: First submitted 2016-01-13; First posted 2017-05-12 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Urinary Tract Infections (UTI's)
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Applicator with LACTIN-V Treatment (Active Comparator): Vaginal applicator containing Lactobacillus crispatus CTV-05
  Interventions: Drug: Lactobacillus crispatus CTV-05
- Applicator with Placebo (Placebo Comparator): Inactive vaginal applicator without any drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus crispatus CTV-05 — vaginal applicator with medium containing drug
  Other Names: Lactin-V
  Arms: Applicator with LACTIN-V Treatment
Drug: Placebo — vaginal applicator with medium containing no drug
  Arms: Applicator with Placebo

SUMMARY:
The purpose of this research is to see whether LACTIN-V (Lactobacillus crispatus CTV-05) is an effective method of preventing recurrent urinary tract infections (UTI's) and to learn the side effects of LACTIN-V. LACTIN-V is a vaginal applicator that contains Lactobacillus crispatus, an organism found naturally in the vaginas of healthy women. Lactobacillus bacteria are thought to help prevent other bacteria such as E. coli from causing UTI's. This is a double blind study comparing active product to a placebo (inactive vaginal applicator without any medicine).

DETAILED DESCRIPTION:
The initial study visit will take about one hour. Participants will read, discuss and sign a consent form. Investigators will have the patient collect a mid-stream urine sample which will be sent to the research lab to confirm the participant has a urinary tract infection (UTI). Participants will than be given Macrobid twice a day for five days for UTI treatment. If the results of the screening show eligibility for this study, investigators will ask the participant to return to the clinic within 3-10 day after completing UTI treatment for a randomization visit (v1).

Visit 1 (Randomization Visit):

During this visit, the participant will be asked about any urinary or vaginal symptoms. The participant will be asked to provide a urine sample to see if the UTI has resolved and for a pregnancy test. The participant will have a physical exam including a pelvic and speculum exam. A study nurse practitioner will collect vaginal specimens to test for vaginal bacteria and vaginal infections.

Next, the participant will be randomly assigned (like flipping a coin) to use LACTIN-V or placebo vaginal applicators. The participant will not be told which product is being used, and the researchers will not know until the end of the study. The participant will not be able to tell which one is being used. Each LACTIN-V applicator contains Lactobacillus crispatus CTV-O5 and other preservatives. Each placebo suppository contains other preservatives.

Participants will be instructed how to use the applicators. The participant will also be given written instructions on how to use, store, and handle the applicators, and a diary to record when the participant uses the applicators and any symptoms that may happen during the study. (Participants will be given 15 applicators).The participant will insert 15 applicators during this study. The applicators are to be used daily for five days during the first week and then once per week for 10 weeks starting the second week. To insert an applicator, the participant will hold one applicator between a thumb and finger (like a tampon),insert the applicator into the opening of the vagina, and then push the applicator plunger. The participant will insert the first applicator in the clinic during this visit. The participant will be asked not to have sexual intercourse or use tampons for 24 hours after inserting an applicator. The participant will also be asked not to use spermicidal vaginal products. The participant will also be asked not to use other vaginal products such as creams, gels, foams, sponges, lubricants, or douches or take antibiotics for a UTI during this study unless the participants doctor prescribes it. The visit will take 30-60 minutes.

Visits 2-6 The participant will then be asked to return to the Hall Health clinic in 2 weeks and then once a month for the next 4 months, after the randomization visit. During these visits a study nurse practitioner will ask about any side-effects that may have occurred from the study drug or placebo. The study nurse practitioner will also ask if the participant had any UTI's since the last visit. The participant will be asked to give a urine sample for culture. The participant will also have a physical exam, and vaginal tests for infection, lactobacillus (including lactobacillus from LACTIN-V) and E. coli. A speculum exam will only be done at v1 and the last visit unless the participant has symptoms of a vaginal infection. The last visit will include a urine pregnancy test. These visits will take 30 minutes.

Other Visits:

If the participant has a UTI or vaginal infection during the study, the participant will be seen at Hall Health for treatment. The participant will be treated with a standard medication at no cost.. If a UTI occurs during the study the participant will continue to use the study applicator on schedule.

ELIGIBILITY:
Inclusion Criteria:

* pre-menopausal women
* present with an acute, uncomplicated, culture confirmed UTI, defined as dysuria, urgency and/or frequency
* at least one previous medically diagnosed UTI in past 12 months
* using a reliable method of birth control ie: history of tubal ligation, male partner with vasectomy, steroidal contraception, Nuva-Ring, IUD, use of non spermicidal condoms or abstinence.
* can provide written consent
* can understand and read English

Exclusion Criteria:

* history of urogenital infection within the past 30 days, including: UTI, medically diagnosed vaginitis
* current symptoms suggestive of pyelonephritis (fever>100.4, flank pain of costovertebral angle tenderness, nausea and vomiting
* history of functional or anatomic urologic abnormalities, urologic surgery of chronic urinary catheterization
* history of pyelonephritis within the past 6 months
* diagnosis of N. gonorrhoeae, C. trachomatis or T. vaginalis on two or more occasions during previous six months
* known HIV infection of seropositivity
* investigational drug use within 30 days of enrollment visit or current participation in another clinical trial
* diabetes, other significant medical problem or intercurrent acute illness that in the Nurse Practitioner's and/or Principal Investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objective.

At the randomization visit, has any of the following findings on pelvic or other physical examination:

* unable to visualize cervix
* clinically significant abnormalities, such as inflammation, erosion and/or petechiae (bleeding under the skin) of external genitalia, vaginal or cervix on visual examination
* clinically significant tenderness on bimanual examination during the pelvic examination
* evidence of vaginitis or a sexually-transmitted disease
* any diagnosis requiring antibiotics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann E Stapleton, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Hall Health Primary Care Center, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Applicator With LACTIN-V Treatment | Applicator With Placebo
Started | 14 | 13
Completed | 12 | 12
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Applicator With LACTIN-V Treatment | Applicator With Placebo | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: UTI Incidence as Described Below, Over the 16 Week Study Period Following Randomization, in the LACTIN-V Treatment Group (Group A) as Compared to the Placebo Group (Group B).
Description: Symptomatic UTI : Comparison of the number (%) of subjects over the 16-week study period following randomization, with at least one symptomatic UTI (as defined above) in the 2 intervention groups
Time Frame: Week 2-18
Population: completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Applicator With LACTIN-V Treatment | Applicator With Placebo
Number analyzed (Participants) | 12 | 12
Participants | 7 | 7

2. Secondary Outcome: Parameter of Vaginal Colonization
Description: Lactobacillus crispatus positive (as assessed by repPCR) at Weeks 0,2,6,10,14, and 18 in the Lactin-V group as compared to the placebo group
Time Frame: Weeks 0, 2, 6, 10, 14 and18
Measure: Number; unit: Number of Participants with Lactobac
Arm/Group | Applicator With LACTIN-V Treatment | Applicator With Placebo
Number analyzed (Participants) | 12 | 12
Number of Participants with Lactobac
  Week 0 | 0 | 0
  Week 2 | 7 | 0
  Week 6 | 8 | 0
  Week 10 | 9 | 0
  Week 14 | 9 | 0
  Week 18 | 7 | 0

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Applicator With LACTIN-V Treatment | Applicator With Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 14/14 | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Applicator With LACTIN-V Treatment (N=14) | Applicator With Placebo (N=13)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 | 0
Eye disorders (Eye disorders) | 0 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 4 | 4
Infections and Infestations (Infections and infestations) | 7 | 6
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 0
Nervous system disorders (Nervous system disorders) | 5 | 2
Renal and urinary disorders (Renal and urinary disorders) | 5 | 7
Reproductive system and breast disorders (Reproductive system and breast disorders) | 7 | 7
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-02-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03151967/Prot_SAP_000.pdf
  • Informed Consent Form (2015-04-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT03151967/ICF_001.pdf